CLINICAL TRIAL: NCT00523614
Title: Use of OCs Containing Dienogest and Risk of Venous Thromboembolism
Brief Title: Use of Oral Contraceptives (OCs) Containing Dienogest and Risk of Venous Thromboembolism
Status: Completed | Type: Observational
Sponsor: Center for Epidemiology and Health Research, Germany (Other)
Collaborators: Bayer (Industry)
Responsible Party: Juergen C Dinger, MD, PhD, Principal Investigator, Center for Epidemiology and Health Research, Germany
Other Study IDs: ZEG2007_02
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Results first posted 2009-12-02 (Estimated); Last update posted 2010-03-23 (Estimated); Status verified 2010-03

CONDITIONS: Venous Thromboembolism
Keywords: venous thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Cases
- 2: Controls

SUMMARY:
The objective of this study is to compare the risk of venous thromboembolism (VTE) of oral contraceptives with non-use, focusing specifically on Valette® compared to other users of low estrogen dose combined oral contraceptives.

DETAILED DESCRIPTION:
This is a population-based case-control study in Germany.

Cases are women who are between 15 and 49 years old with a diagnosis of venous thromboembolism (VTE). The VTE is diagnosed in Germany between January 2002 und December 2007.

Controls are women who are between 15 and 49 years old without a VTE diagnosis. About 4 controls matched by year of birth and region will be allocated to each case.

Both cases and controls will receive a similar self-administered questionnaire except of some case-specific questions which are not applicable for the controls.

Study participants will be asked for their informed consent. Data confidentiality will be ensured by the Berlin Center for Epidemiology and Health Research.

ELIGIBILITY:
Inclusion Criteria:

* cases: women with a venous thromboembolism who are between 15 and 49 years old
* control: women without a venous thromboembolism diagnosis who are between 15 and 49 years old

Exclusion Criteria:

* women outside the defined age range
* women with severe language problems
* women who are not willing to participate

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cases: women between 15 and 49 years old with a VTE diagnosed in Germany between 2002 and 2007
  Controls: population sample
Sampling Method: Non-Probability Sample
Enrollment: 3400 (Actual)
Dates: Start 2007-07; Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juergen C Dinger, MD, PhD, Principal Investigator — Center for Epidemiology and Health Research
Locations (1):
- Center for Epidemilogy and Health Research, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Identification started in spring 2007 and ended in January 2008. Cases (VTE=venous thromboembolism diagnosed in Germany between 01/2002 and 01/2008) were identified by primary care physicians. For each case 4 community-based controls (no VTE between 01/2002 and 01/2008) were selected.The controls were identified from randomly selected households.
Groups:
- Cases: Women with a venous thromboembolism who are between 15 and 49 years old
- Controls: Women without a venous thromboembolism diagnosis who are between 15 and 49 years old
Period: Overall Study
Arm/Group | Cases | Controls
Started | 680 (As this is a case-control study the categories "started" and "completed" are not really applicable.) | 2720 (As this is a case-control study the categories "started" and "completed" are not really applicable.)
Completed | 680 (As this is a case-control study the categories "started" and "completed" are not really applicable.) | 2720 (As this is a case-control study the categories "started" and "completed" are not really applicable.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cases | Controls | Total
Number analyzed (Participants) | 680 | 2720 | 3400
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 60 | 75
  Between 18 and 65 years | 665 | 2660 | 3325
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 36.1 (9.0) | 36.1 (9.0) | 36.1 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 680 | 2720 | 3400
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 680 | 2720 | 3400

OUTCOME MEASURES:

1. Primary Outcome: Risk of Venous Thromboembolism (VTE) Between Women Who Use Dienogest/Ethinylestradiol (DNG/EE) and Women Who Use Other Low-dose Combined Oral Contraceptives (COC)
Description: The time frame is the time when venous thromboembolism (VTE) was diagnosed in the cases group. VTE includes deep venous thrombosis and pulmonary embolism. These clinical endpoints were established by magnetic resonance imaging, spiral computer tomography, duplex sonography, and lung scintigraphy.
Time Frame: 01/2002 - 01/2008
Measure: Number; unit: Participants
Groups:
- Controls: Women without a venous thromboembolism who are between 15 and 49 years old
Arm/Group | Cases | Controls
Number analyzed (Participants) | 680 | 2720
Participants
  Exposed DNG/EE COC | 35 | 106
  Exposed low-dose COC | 161 | 423
Statistical Analysis 1: Comparison: Cases vs Controls; Null hypothesis: OR ≥ 2 (VTE of DNG/EE vs. other low-dose COC); Test type: Non-Inferiority or Equivalence — Size of the study adapted to the use of DNG/EE in female fertile age. Market share of DNG/EE of 13% in Germany. Assuming that 30% of women in the fertile age range were current users of OCs, a prevalence of current use of DNG/EE of about 4% was estimated. Based on these data the number of cases needed to exclude a twofold increased VTE risk was estimated at about 500-700 cases (based on four controls per case); p < 0.05, Regression, Logistic; Odds Ratio (OR) = 0.89, 95% CI [0.57 to 1.39]

ADVERSE EVENTS:
Arm/Group | Cases | Controls
Serious Adverse Events (participants affected / at risk) | 0/680 | 0/2720
Other Adverse Events (participants affected / at risk) | 0/680 | 0/2720

LIMITATIONS AND CAVEATS:
This is an observational study. The possibility of bias and residual confounding cannot be entirely eliminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes